CLINICAL TRIAL: NCT00944866
Title: Effects of Cox-II Inhibitor on Biochemical Markers in Cardiovascular-related Adverse Effects
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Chung Hsing University (Other)
Responsible Party: En-Pei Isabel Chiang, National Chung Hsing University
Other Study IDs: C07146
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- RA with drug
- RA without drug

SUMMARY:
The selective cyclooxygenase-2 (COX-2) inhibitors have been associated with increased cardiovascular risk. The goal of the present study is to investigate the impacts of COX-2 inhibitors on biochemical indices in cardiovascular disease. As the reviewer suggested, the investigators propose to study the effects of Cox-II inhibitor using experimentally induced hyperlipidemic rats. Plasma total cholesterol, LDL and triglyceride concentrations will be determined before and after animals treated with cyclooxygenase-2 (COX-2) inhibitors. Biochemical markers related to cardiovascular events including prostaglandin I2, thromboxaneA2 and others will also be investigated. The investigators will also investigate these biochemical markers in patients taking Celecoxib and NSAIDs. The investigators hope these studies will reveal clinically useful biochemical markers for cardiovascular events in patients taking Cox-II inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Male/female age >18
* Clinical diagnosed of arthritis

Exclusion Criteria:

* Must not be pregnant/breastfeeding
* Other conditions may lead to exclusion from the trial (e.g. Diabetes mellitus, malignant melanoma, cardiac conduction disorders, hepatic/renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Arthritis
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

REFERENCES:
- [Derived] Chang HY, Tang FY, Chen DY, Chih HM, Huang ST, Cheng HD, Lan JL, Chiang EP. Clinical use of cyclooxygenase inhibitors impairs vitamin B-6 metabolism. Am J Clin Nutr. 2013 Dec;98(6):1440-9. doi: 10.3945/ajcn.113.064477. Epub 2013 Oct 23. PMID 24153347